CLINICAL TRIAL: NCT07067268
Title: A Multicenter, Randomized Controlled, Phase II Trail of Tislelizumab Combined With Capecitabine for Nasopharyngeal Carcinoma Patients With Residual Epstein-Barr Virus (EBV) DNA After Radiotherapy
Brief Title: Tislelizumab Combined With Capecitabine for Nasopharyngeal Carcinoma With Residual EBV DNA After Radiotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chaosu Hu, Professor, M.D., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BioNPC-03
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: Nasopharyngeal Carcinoma; EBV DNA; Tislelizumab; capecitabine; Adjuvant therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant therapy arm (Experimental): Tislelizumab combined with capecitabine therapy
  Interventions: Drug: Adjuvant therapy
- Control arm (No Intervention): Clinical follow-up and surveillance only

INTERVENTIONS:
Drug: Adjuvant therapy — Tislelizumab: 200 mg IV on day 1, every 3 weeks Capecitabine: 1000 mg/m² orally twice daily on days 1-14，every 3 weeks Treatment duration: 8 cycles
  Arms: Adjuvant therapy arm

SUMMARY:
This study aims to explore the efficacy and safety of tislelizumab combined with capecitabine in nasopharyngeal carcinoma patients with residual plasma EBV DNA after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Histologically confirmed nasopharyngeal carcinoma;
3. Expected survival time ≥12 weeks;
4. ECOG performance status: 0-1;
5. Received definitive radiotherapy (± induction and/or concurrent chemotherapy);
6. Plasma EBV DNA >0 copies/mL within the period from 1 week before to 4 weeks after completion of radiotherapy ;
7. Adequate organ function meeting the following criteria: Hematological: a. Hemoglobin (HB) ≥90 g/L; b. Absolute neutrophil count (ANC) ≥1.0×10⁹/L; c. Platelet count (PLT) ≥80×10⁹/L; Biochemical: a. Total bilirubin (BIL) <1.5× upper limit of normal (ULN); b. ALT and AST <2.5×ULN; c. Serum creatinine (Cr) ≤ULN, and creatinine clearance rate ≥50 mL/min (calculated by Cockcroft-Gault formula); d. Normal myocardial enzymes and thyroid function; e. Normal cardiac function assessed by echocardiography.
8. Signed informed consent with willingness to comply with the study protocol.

Exclusion Criteria:

1. Histologically confirmed keratinizing squamous cell carcinoma (WHO I)；
2. Distant metastasis detected by pre-treatment clinical or imaging examinations;
3. History of allergy to any component of monoclonal antibodies, tislelizumab, or capecitabine;
4. History of autoimmune diseases, except for the following conditions (eligible after evaluation):

   1. Autoimmune-related hypothyroidism on stable thyroid hormone replacement therapy;
   2. Type I diabetes mellitus under stable insulin therapy with controlled blood glucose;
5. Previous or concurrent malignancies (except those cured and disease-free for >5 years, e.g., basal cell carcinoma, cervical carcinoma in situ);
6. Positive pregnancy test in women of childbearing potential;
7. Concurrent medical conditions that may compromise patient enrollment or safety during the study;
8. History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, organizing pneumonia, idiopathic pneumonia, or other active pulmonary diseases;
9. Active psychiatric disorders or other mental conditions affecting informed consent comprehension;
10. Uncontrolled active infections, including tuberculosis, hepatitis B (HBsAg+), hepatitis C, or HIV (HIV antibody+);
11. Significant cardiovascular diseases: NYHA Class II or higher, myocardial infarction within 1 year, unstable angina, or supraventricular/ventricular arrhythmias requiring clinical intervention;
12. Factors affecting drug administration, distribution, metabolism, or excretion (e.g., psychiatric/neurological disorders, chronic diarrhea, ascites, pleural effusion);
13. Unwillingness to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  Defined from date of randomization to date of first documentation of progression or death due to any cause

SECONDARY OUTCOMES:
Overall survival | 3 years
  The time from enrollment to death due to any cause or censored at the date of last follow-up.
Toxicities | 3 years
  Adverse effects (AE) are evaluated by CTCAE 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Universtiy Shanghai Cancer Centre, Shanghai, China, China